CLINICAL TRIAL: NCT00570102
Title: Trial to Reduce IDDM in the Genetically at Risk (TRIGR): the Pilot Study
Brief Title: Nutritional Prevention Pilot Trial for Type 1 Diabetes
Acronym: MIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Academy of Finland (Other); European Union (Other); Juvenile Diabetes Research Foundation (Other); Diabetes Research Foundation, Finland (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Mikael Knip, Professor of Pediatrics, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 195003; BHM4-CT96-0233
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: dietary manipulation; infants; feasibility; Type 1 Diabetes Mellitus, Beta-cell Autoimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A highly hydrolyzed casein formula (Active Comparator)
  Interventions: Dietary Supplement: A highly hydrolyzed formula
- A conventiona cow's milk based formula (Placebo Comparator)
  Interventions: Dietary Supplement: A regular cow's milk based formula

INTERVENTIONS:
Dietary Supplement: A highly hydrolyzed formula — Weaning to a highly hydrolyzed formula, avoidance of all supplemental food containing cow's milk proteins and/or bovine serum albumin up to the age of 6-8 months
  Arms: A highly hydrolyzed casein formula
Dietary Supplement: A regular cow's milk based formula — Weaning to a regular cow's milk based formula supplemented with 20% of the highly hydrolyzed formula used in arm 1 to make the study formulas similar in smell and taste, avoidance of all supplemental food containing cow's milk proteins and/or bovine serum albumin
  Arms: A conventiona cow's milk based formula

SUMMARY:
The overall objective of the study is to assess whether complete avoidance of cow's milk (CM) proteins, for at least the first 6 months of life, prevents type 1 diabetes (insulin-dependent diabetes mellitus, IDDM) in genetically susceptible children who have a mother, biological father or sibling affected by type 1 diabetes.

DETAILED DESCRIPTION:
Among the environmental factors leading to type 1 diabetes in childhood, the most important are certain viral infections and possibly some dietary factors. Among the latter cow's milk proteins are of special interest. They have been shown to be involved in the pancreatic beta-cell lesion in animal experiments. In humans there are some indications of a role of early exposure to cow's milk proteins as a risk factor for later type 1 diabetes. The hypothesis has not been confirmed, but a randomized, controlled double-blinded intervention trial should provide a definite answer.

This study aims at assessing whether one can decrease the future incidence of beta-cell autoimmunity and/or type 1 diabetes in children who have an increased genetic risk for the disease, by administering in infancy after breast feeding until the age of 6-8 months such a formula, in which the cow's milk proteins have been hydrolyzed to smaller peptides. The children in the control group, carrying a similar increased genetic risk, will receive a conventional cow's milk based formula .

This project is a pilot multicenter trial comprising 15 hospitals in Finland.

ELIGIBILITY:
Inclusion Criteria:

* the participant must have a mother, biological father or sibling with type 1 diabetes
* the participant must carry a susceptible HLA genotype(HLA-DQB1*02 and/or DQB1*0302 without protective alleles (DQB1*0301, *0602 and *0603)

Exclusion Criteria:

* no telephone
* no accessibility to any of the research centers
* inability of parents to understand the study and instructions
* unwillingness/inability to feed the infant CM-containing food for any reason (e.g. religious, cultural reasons)
* gestational age less than 36 weeks
* Any severe illness such as chromosomal abnormalities, congenital malformations, respiratory failure, enzyme deficiencies of the newborn.
* the newborn infant has received any cow's milk-based product prior to randomization

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 1995-02; Primary Completion 2004-03 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Positivity for two or more diabetes-associated autoantibodies and/or clinical type 1 diabetes | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans K Åkerlom, MD, PhD, Principal Investigator — University of Helsinki, Helsinki, Finland
Locations (18):
- Finland (18):
  - Jorvi Hospital, Espoo
  - Kanta-Häme Central Hospital, Department of Pediatrics, Hämeenlinna
  - University of Helsinki, Department of Obstetrics and Gynecology, Helsinki
  - National Public Health Institute, Helsinki
  - Helsinki University Hospital, Maternity Hospital, Helsinki
  - University of Helsinki, Hospital for Children and Adolescents, Helsinki
  - North Karelia Central Hospital, Joensuu
  - Central Finland Central Hospital, Jyväskylä
  - Kymenlaakso Central Hospital, Department of Pediatrics, Kotka
  - University of Kuopio, Department of Pediatrics, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - South Karelia Central Hospital, Lappeenranta
  - University of Oulu, Department of Pediatrics, Oulu
  - Satakunta Central Hospital, Pori
  - South Ostrobothnia Central Hospital, Seinäjoki
  - Tampere University Hospital, Department of Pediatrics, Tampere
  - University of Turku, Department of Virology, Turku
  - Vaasa Central Hospital, Vaasa

REFERENCES:
- [Background] Akerblom HK, Savilahti E, Saukkonen TT, Paganus A, Virtanen SM, Teramo K, Knip M, Ilonen J, Reijonen H, Karjalainen J, et al. The case for elimination of cow's milk in early infancy in the prevention of type 1 diabetes: the Finnish experience. Diabetes Metab Rev. 1993 Dec;9(4):269-78. doi: 10.1002/dmr.5610090407. No abstract available. PMID 7924824
- [Background] Akerblom HK, Knip M. Putative environmental factors in Type 1 diabetes. Diabetes Metab Rev. 1998 Mar;14(1):31-67. doi: 10.1002/(sici)1099-0895(199803)14:13.0.co;2-a. PMID 9605629
- [Background] Knip M, Akerblom HK. IDDM prevention trials in progress--a critical assessment. J Pediatr Endocrinol Metab. 1998 Apr;11 Suppl 2:371-7. No abstract available. PMID 9642667
- [Background] Knip M, Akerblom HK. Environmental factors in the pathogenesis of type 1 diabetes mellitus. Exp Clin Endocrinol Diabetes. 1999;107 Suppl 3:S93-100. doi: 10.1055/s-0029-1212160. PMID 10522815
- [Background] Vaarala O, Hyoty H, Akerblom HK. Environmental factors in the aetiology of childhood diabetes. Diabetes Nutr Metab. 1999 Apr;12(2):75-85. No abstract available. PMID 10554890
- [Background] Akerblom HK, Vaarala O, Hyoty H, Ilonen J, Knip M. Environmental factors in the etiology of type 1 diabetes. Am J Med Genet. 2002 May 30;115(1):18-29. doi: 10.1002/ajmg.10340. PMID 12116173
- [Background] Knip M, Akerblom HK. Early nutrition and later diabetes risk. Adv Exp Med Biol. 2005;569:142-50. doi: 10.1007/1-4020-3535-7_21. PMID 16137119
- [Background] Knip M, Veijola R, Virtanen SM, Hyoty H, Vaarala O, Akerblom HK. Environmental triggers and determinants of type 1 diabetes. Diabetes. 2005 Dec;54 Suppl 2:S125-36. doi: 10.2337/diabetes.54.suppl_2.s125. PMID 16306330
- [Result] Paronen J, Knip M, Savilahti E, Virtanen SM, Ilonen J, Akerblom HK, Vaarala O. Effect of cow's milk exposure and maternal type 1 diabetes on cellular and humoral immunization to dietary insulin in infants at genetic risk for type 1 diabetes. Finnish Trial to Reduce IDDM in the Genetically at Risk Study Group. Diabetes. 2000 Oct;49(10):1657-65. doi: 10.2337/diabetes.49.10.1657. PMID 11016449
- [Result] Hamalainen AM, Ronkainen MS, Akerblom HK, Knip M. Postnatal elimination of transplacentally acquired disease-associated antibodies in infants born to families with type 1 diabetes. The Finnish TRIGR Study Group. Trial to Reduce IDDM in the Genetically at Risk. J Clin Endocrinol Metab. 2000 Nov;85(11):4249-53. doi: 10.1210/jcem.85.11.6987. PMID 11095462
- [Result] Ronkainen MS, Hamalainen AM, Koskela P, Akerblom HK, Knip M; Finnish Trigr Study Group. Pregnancy induces nonimmunoglobulin insulin-binding activity in both maternal and cord blood serum. Clin Exp Immunol. 2001 May;124(2):190-6. doi: 10.1046/j.1365-2249.2001.01506.x. PMID 11422194
- [Result] Hamalainen AM, Savola K, Kulmala PK, Koskela P, Akerblom HK, Knip M; Finnish TRIGR Study Group. Disease-associated autoantibodies during pregnancy and at birth in families affected by type 1 diabetes. Clin Exp Immunol. 2001 Nov;126(2):230-5. doi: 10.1046/j.1365-2249.2001.01676.x. PMID 11703365
- [Result] Sadeharju K, Hamalainen AM, Knip M, Lonnrot M, Koskela P, Virtanen SM, Ilonen J, Akerblom HK, Hyoty H; Finnish TRIGR Study Group. Enterovirus infections as a risk factor for type I diabetes: virus analyses in a dietary intervention trial. Clin Exp Immunol. 2003 May;132(2):271-7. doi: 10.1046/j.1365-2249.2003.02147.x. PMID 12699416
- [Result] Akerblom HK, Virtanen SM, Ilonen J, Savilahti E, Vaarala O, Reunanen A, Teramo K, Hamalainen AM, Paronen J, Riikjarv MA, Ormisson A, Ludvigsson J, Dosch HM, Hakulinen T, Knip M; National TRIGR Study Groups. Dietary manipulation of beta cell autoimmunity in infants at increased risk of type 1 diabetes: a pilot study. Diabetologia. 2005 May;48(5):829-37. doi: 10.1007/s00125-005-1733-3. Epub 2005 Apr 19. PMID 15838685
- [Result] Tiittanen M, Paronen J, Savilahti E, Virtanen SM, Ilonen J, Knip M, Akerblom HK, Vaarala O; Finnish TRIGR Study Group. Dietary insulin as an immunogen and tolerogen. Pediatr Allergy Immunol. 2006 Nov;17(7):538-43. doi: 10.1111/j.1399-3038.2006.00447.x. PMID 17014631
- [Result] Sadeharju K, Knip M, Virtanen SM, Savilahti E, Tauriainen S, Koskela P, Akerblom HK, Hyoty H; Finnish TRIGR Study Group. Maternal antibodies in breast milk protect the child from enterovirus infections. Pediatrics. 2007 May;119(5):941-6. doi: 10.1542/peds.2006-0780. PMID 17473095
- [Result] Knip M, Virtanen SM, Seppa K, Ilonen J, Savilahti E, Vaarala O, Reunanen A, Teramo K, Hamalainen AM, Paronen J, Dosch HM, Hakulinen T, Akerblom HK; Finnish TRIGR Study Group. Dietary intervention in infancy and later signs of beta-cell autoimmunity. N Engl J Med. 2010 Nov 11;363(20):1900-8. doi: 10.1056/NEJMoa1004809. PMID 21067382
- [Derived] Hyytinen M, Savilahti E, Virtanen SM, Harkonen T, Ilonen J, Luopajarvi K, Uibo R, Vaarala O, Akerblom HK, Knip M; Finnish TRIGR Pilot Study Group. Avoidance of Cow's Milk-Based Formula for At-Risk Infants Does Not Reduce Development of Celiac Disease: A Randomized Controlled Trial. Gastroenterology. 2017 Oct;153(4):961-970.e3. doi: 10.1053/j.gastro.2017.06.049. Epub 2017 Jul 5. PMID 28687275
- [Derived] de Goffau MC, Luopajarvi K, Knip M, Ilonen J, Ruohtula T, Harkonen T, Orivuori L, Hakala S, Welling GW, Harmsen HJ, Vaarala O. Fecal microbiota composition differs between children with beta-cell autoimmunity and those without. Diabetes. 2013 Apr;62(4):1238-44. doi: 10.2337/db12-0526. Epub 2012 Dec 28. PMID 23274889
- See also: The TRIGR Study proper tests the hypothesis whether weaning to a highly hydrolyzed formula reduces the cumulative incidence of beta-cell autoimmunity and clinical diabetes in subjects with increased genetic disease susceptibility — http://trigr.epi.usf.edu